CLINICAL TRIAL: NCT07046273
Title: A Multicenter, Randomized, Open, Parallel-controlled, Phase III Clinical Study on the Efficacy and Safety of Semaglutide and Ozempic® in Patients With Type 2 Diabetes
Brief Title: Phase III Clinical Study on the Efficacy and Safety of Semaglutide and Ozempic® in Patients With Type 2 Diabetes
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTP-F027-002
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F027 (Experimental): The starting dose is 0.25 mg once weekly. After 4 weeks the dose should be increased to 0.5 mg once weekly. After at least 4 weeks with a dose of 0.5 mg once weekly, the dose can be increased to 1 mg once weekly for 24 weeks.
  Interventions: Drug: F027
- Ozempic® (Active Comparator): The starting dose is 0.25 mg once weekly. After 4 weeks the dose should be increased to 0.5 mg once weekly. After at least 4 weeks with a dose of 0.5 mg once weekly, the dose can be increased to 1 mg once weekly for 24 weeks.
  Interventions: Drug: Ozempic®

INTERVENTIONS:
Drug: F027 — The starting dose is 0.25 mg once weekly. After 4 weeks the dose should be increased to 0.5 mg once weekly. After at least 4 weeks with a dose of 0.5 mg once weekly, the dose can be increased to 1 mg once weekly for 24 weeks.
  Arms: F027
Drug: Ozempic® — The starting dose is 0.25 mg once weekly. After 4 weeks the dose should be increased to 0.5 mg once weekly. After at least 4 weeks with a dose of 0.5 mg once weekly, the dose can be increased to 1 mg once weekly for 24 weeks.
  Arms: Ozempic®

SUMMARY:
This study is a multicenter, randomized, open, parallel-controlled, Phase III clinical study aimed to evaluate the efficacy and safety of semaglutide injection and Ozempic® in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 1) Voluntary signing of informed consent; 2) Aged 18-75 years (inclusive) at the time of signing the informed consent, male or female; 3) Diagnosed with type 2 diabetes according to the WHO diabetes diagnostic criteria; 4) Laboratory tests at the research center at screening: 7.5%≤HbA1c≤10.5%; 5) Before randomization, study participants received stable doses of metformin (≥1500mg/day or maximum tolerated dose: <1500mg/day, but ≥1000mg/day) for at least 8 weeks (maximum tolerated dose must be supported by previous medical records); 6) Body mass index (BMI) ≥18.5kg/m2 and ≤35.0kg/m2 at screening; 7) Willing and able to undergo treatment and follow-up as required by the protocol.

Exclusion Criteria:

1. Type 1 diabetes, special type of diabetes;
2. Received hypoglycemic drugs other than metformin (including Chinese medicine) within 8 weeks before randomization;
3. Used non-diabetes treatment drugs that may have a significant impact on glucose metabolism for 1 week or more within 3 months before randomization, such as glucocorticoids (systemic glucocorticoids used for <7 days, excluding inhalation, ocular medication or topical application), sympathetic nerve stimulants (such as isoproterenol, dopamine, atropine, etc.), growth hormone, high-dose salicylates (300 mg/day and above), danazol, octreotide and anabolic androgenic steroids (such as oxymetholone, oxandrolone, etc.);
4. Has a history of ≥2 episodes of grade 3 hypoglycemia within 1 year before randomization;
5. Diabetic ketoacidosis or hyperglycemic hyperosmolar state within 3 months before randomization;
6. Severe complications of diabetes at screening: such as proliferative diabetic retinopathy, macular edema; history of renal transplantation; severe peripheral vascular disease (such as amputation, chronic foot ulcers, intermittent claudication);
7. Untreated or poorly controlled hypertension (defined as systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg) at screening/randomization;
8. Cardiovascular diseases such as acute coronary syndrome (including but not limited to acute myocardial infarction, or unstable angina), arrhythmia requiring treatment, severe heart failure (refer to New York Heart Association heart function grade III or IV), coronary artery bypass grafting or coronary stent implantation within 6 months before screening;
9. New cerebrovascular accident (including ischemic stroke, hemorrhagic stroke and transient ischemic attack, etc.) within 6 months before screening;
10. Severe trauma or severe infection or surgery that may affect blood sugar control within 1 month before screening;
11. History of acute or chronic pancreatitis;
12. History of cholecystitis due to cholelithiasis or other reasons within 6 months before screening;
13. Cushing's syndrome, hyperthyroidism, and uncontrolled hypothyroidism at screening;
14. Significant gastric emptying abnormalities (such as gastric outlet obstruction) and severe gastrointestinal diseases at screening;
15. Any disease that may cause hemolysis or red blood cell instability and affect HbA1c detection, such as blood system tumors, hemolytic anemia, sickle cell disease;
16. History or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2);
17. History of malignant tumors in the past 5 years (regardless of organ system, whether treated or not, and whether there is evidence of recurrence or metastasis) or currently being evaluated for potential malignant tumors, but excluding clinically cured cervical carcinoma in situ and skin basal cell carcinoma;
18. Meet any of the following criteria at screening:

    Liver function impairment: ALT or AST ≥ 5 times the upper limit of normal, or total bilirubin ≥ 2 times the upper limit of normal; Renal function impairment: glomerular filtration rate (eGFR, CKD-EPI formula) < 45mL/min/1.73m2; Fasting triglyceride (TG) ≥ 5.7mmol/L after stable medication; Calcitonin ≥ 50ng/L; Hemoglobin ≤ 100g/L; Thyrotropin (TSH) > 6mIU/L after stable medication; Blood amylase or lipase ≥ 3 times the upper limit of normal; Hepatitis C virus antibody, human immunodeficiency virus antibody, syphilis serological test results are positive, hepatitis B virus surface antigen is positive and HBV-DNA is positive.
19. Known allergy to any component of semaglutide injection or allergy to other GLP-1 RA drugs;
20. Donated blood or lost ≥400mL of blood within 3 months before screening, or received blood transfusion therapy, or planned to donate blood during the trial;
21. Received other clinical research drugs or device treatments within 3 months before screening, or participated in other drug clinical trials and are still within 5 half-lives of the trial drug, whichever is older; or planned to participate in other clinical studies during the trial;
22. Have a history of drug abuse (including drug abuse) and/or alcohol dependence within 6 months before screening;
23. Mental disorder or language barrier, unable to fully understand and cooperate;
24. Pregnant or lactating women;
25. Male and female research participants who have fertility plans during the trial and within 2 months after the last dose of the trial drug, or are unwilling to take reliable contraceptive measures for contraception;
26. Other situations that the researcher considers unsuitable for participation in this study. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c from baseline | Week 32

SECONDARY OUTCOMES:
Change in HbA1c from baseline | Week 20
Percentage of Participants Who Achieved HbA1c <6.5% | Week 32
Percentage of participants who achieved HbA1c < 7.0% | Week 32
Change in Fasting Glucose | Week 20 ,32
Change in Body Weight | Week 32
Collect the incidence of adverse events (AEs)/serious adverse events (SAEs) through vital signs, physical examination, laboratory tests, 12-lead electrocardiogram, etc. | Week 32
Incidence of hypoglycemic events and acute pancreatitis | Week 32
Incidence of anti-drug antibodies (ADA) and neutralizing antibodies (Nab) | Week 32
Semaglutide steady-state trough concentration (Css, min) | Week 32

IPD SHARING:
Plan to Share IPD: Undecided